CLINICAL TRIAL: NCT03343730
Title: Diabetic Retinopathy Screening With Non-mydriatic Color Fundus Camera in the Primary Care Clinic
Brief Title: RetinaVue Diabetic Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, James Dalton, Attending Physician - Primary Care, Bassett Healthcare
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 2078
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Non-mydriatic color fundus photography (Experimental): All participants will receive Non-mydriatic color fundus photography with the RetinaVue camera at an already scheduled annual physical exam or follow up clinic visit with their primary care provider (PCP).
  Interventions: Diagnostic Test: Non-mydriatic color fundus photography with the RetinaVue camera
- Standard of Care (Control) (Active Comparator): All patients will also receive a referral for a dilated eye exam with an eye care professional. A yearly dilated exam as referred by the PCP.
  Interventions: Diagnostic Test: Referral for dilated eye exam with an eye care professional

INTERVENTIONS:
Diagnostic Test: Non-mydriatic color fundus photography with the RetinaVue camera — This hand-held device allows the primary care physician to capture an image of the patient's retina and transmit the image to a board-certified ophthalmologist for interpretation.
  Arms: Non-mydriatic color fundus photography
Diagnostic Test: Referral for dilated eye exam with an eye care professional — All patients will be given a referral to an eye care professional for a routine, dilated, diabetic eye exam.
  Arms: Standard of Care (Control)

SUMMARY:
the purpose of this study is to examine whether the deployment of a non-mydriatic color fundus camera in a rural prime care setting is feasible and improves the detection rate of diabetic retinopathy in patients where adherence rates with recommended ophthalmology screening is low.

DETAILED DESCRIPTION:
The Centers for Disease Control and Prevention (CDC) have estimated that 25.6 million Americans aged 20 years or older have either been diagnosed or undiagnosed with diabetes mellitus. As such, it is crucial for patients to receive routine eye exams during their annual health assessment or diabetes follow-up visit with their primary care physician to check for diabetic retinopathy (DR). Of those Type 2 patients with a known duration of diabetes of less than 5 years, DR was diagnosed in 40% of patients taking insulin and 24% of patients not taking insulin. These percentages are especially concerning since data presented by Schoenfeld and colleagues indicates that approximately 35% of Americans with diabetes mellitus do not receive timely and recommended eye care to detect and treat their DR.10 Reasons for noncompliance include transfer to a retinal specialist, limited personal mobility, and insurance. In addition, patients regularly fail to follow-up with their ophthalmologist or optometrist due to the lack of visual symptoms-the lack of symptoms does not exclude the possibility of early diabetic retinopathy. Per the American Diabetes Association (ADA) guidelines, it is recommended that all Type 2 patients receive annual dilated eye exams. These eye exams must be completed by a knowledgeable and experienced eye care professional (i.e. ophthalmologist or optometrist). Early detection of DR and the preventative effects of therapy is an important aspect for long term vision outcomes.

The long-term goal is to improve the detection of diabetic retinopathy through better-quality measures of patient compliance and screening protocols in the prime care clinic. It is hypothesized that in type II diabetic patients without documented retinal pathology, a hand-held non-mydriatic fundus camera is superior to a referred dilated eye exams for the screening and detection of DR.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Type II diabetes without documented diabetic retinopathy

Exclusion Criteria:

1. Documented ocular pathology that may interfere with image acquisition (i.e. high grade cataract)
2. Macular pathology (i.e. macular degeneration, cystoid macular edema, central serous retinopathy)
3. Inability to attain analyzable RetinaVue image due to ocular pathology or other conditions (such as tremors limiting ability to maintain stable head for image)
4. Acute or emergent ocular pathology that requires urgent assessment by an eye care professional as identified by the RetinaVue camera interpretation report
5. Seen within the last 11 months for a diabetic eye exam.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Diabetic Retinopathy Detection | 3 months
  This study will examine the rate of detection of diabetic retinopathy using an in-clinic retinal camera and standard referral to eye care professional for dilated eye exam

CONTACTS AND LOCATIONS:
Overall Officials: james Dalton, MD, Principal Investigator — Bassett Medical Center
Locations (1):
- Bassett Medical Center, Cooperstown, New York, United States